

# Official Title: Desaturation Validation of INVSENSOR00039

Date of Protocol: August 6, 2019

NCT Number: NCT04112784



## **Desaturation Validation of INVSENSOR00039**

| Protocol/Test Procedure Title | Desaturation Validation of INVSENSOR00039 |
|---|---|
| Lead Investigator | Manager, Clinical Trials Masimo Corporation 52 Discovery, Irvine, CA 92618 |
| Other Investigators | |
| Expected Start Date | TBD |
| Expected End Date | TBD |
| IRB | E&I West Coast Board – IRB00007807 |
| Protocol Version Date | TBD |

#### **Protocol Test Abstract:**

This study is designed to compare the accuracy of a noninvasive measurement of oxygen saturation compared to reference values obtained by a laboratory blood gas analyzer. Arterial blood samples will be collected from healthy adult subjects while undergoing a desaturation procedure wherein the concentration of oxygen inhaled is slowly reduced until the subject's arterial oxygen concentration is approximately 70%. The subject will then be returned to breathing room air.

#### **APPROVALS**

| Author | Date | Engineering | Date |
|-------------------|------|---------------|------|
| N/A | N/A | N/A | N/A |
| Quality Assurance | Date | Manufacturing | Date |
| N/A | N/A | N/A | N/A |

R-TP-20068

## **Desaturation Validation of INVSENSOR00039**



#### STATEMENT OF COMPLIANCE

This document is a protocol for a clinical research study sponsored by Masimo Corporation. The study will be conducted in compliance with all stipulations of this protocol, the conditions of IRB approval, 21 CFR Part 50, 21 CFR Part 56, 21 CFR Part 812, ISO-14155, and International Conference on Harmonisation E6 Good Clinical Practice (ICH GCP).

The protocol, informed consent form(s), recruitment materials, and all participant materials will be submitted to the Institutional Review Board (IRB) for review and approval. Approval of both the protocol and the consent form must be obtained before any participant is enrolled. Any amendment to the protocol will require review and approval by the IRB before the changes are implemented to the study.

#### 1. PURPOSE

The objective of this study is to validate the noninvasive oxygen saturation ( $SpO_2$ ) performance of the Masimo noninvasive INVSENSOR00039 sensor against an arterial blood sample analyzed by a laboratory CO-oximeter reference instrument. Data using the noninvasive devices will be collected from healthy volunteers undergoing a desaturation procedure.

This is a nonrandomized single arm study wherein all subjects are enrolled into the experimental arm and receive the INVSENSOR00039 sensor on one or more fingers. Desaturation will be conducted by reducing the concentration of oxygen the study subject breathes in a controlled manner to obtain noninvasive oxygen saturation readings,  $SpO_{2}$ , at various levels. Reference blood samples will be repeatedly collected from the subject and analyzed using a standard laboratory CO-oximeter. The performance of the sensors will be calculated using Accuracy root mean square ( $A_{RMS}$ ) analysis of the  $SpO_2$  values and the reference CO-oximeter values.

## Outcome Measure:

Performance of the sensors will be determined by comparing the noninvasive oxygen saturation measurement  $(SpO_2)$  of the pulse oximeter sensors to the arterial oxygen saturation (SaO2) value obtained from a reference blood sample and calculating the  $A_{RMS}$  value.

#### 2. BACKGROUND

Masimo Corporation develops non-invasive medical technologies. These devices have applications in the operating room, critical care unit, emergency room, emergency transport vehicles, as well as physician's offices.

An invasive blood sample analyzed by a CO-oximeter reference instrument gives the best measure of arterial oxygen concentration as well as other blood solutes, but cannot measure these parameters continuously and requires skin puncture, arterial line placement and subsequent risk of infection, hematoma, and other physiological damage. Masimo SET and Masimo Rainbow technologies allow real-time, non-invasive monitoring of oxygen saturation (and other blood solutes) and has the potential to improve clinical outcomes while reducing the cost of care and risks to both patients and clinicians associated with arterial and venous punctures.

## 2.1. Technology Background

Pulse oximetry is governed by the following principles:

- Oxyhemoglobin (oxygenated blood) and deoxyhemoglobin (non-oxygenated blood) differ in their absorption of red and infrared light (spectrophotometry).
- The amount of arterial blood in tissue changes with arterial pulses (photoplethysmography). Therefore, the amount of light absorbed by the varying quantities of arterial blood changes as well.

R-TP-20068

## Desaturation Validation of INVSENSOR00039





- Light Emitting Diodes (LEDs)
   (2+ wavelengths)
- Detector

## 2.2. Investigational Devices

The investigational Masimo INVSENSOR00039INVSENSOR00039\_is a disposable sensor intended to provide arterial blood saturation values. The INVSENSOR00039 will communicate with the Masimo Rad-97 Pulse CO-Oximeter to display plethysmograph and parameter values.

INVSENSOR00039 sensors are similar to existing Masimo FDA-cleared sensors

## 3. REFERENCE

 ${\tt Consent\ To\ Be\ A\ Research\ Subject\ Desaturation\ Validation\ of\ \ INVSENSOR00039}$ 

Health Assessment Questionnaire Desaturation Validation of INVSENSOR00039

Desaturation Validation of INVSENSOR00039 Recruitment Script

Desaturation Validation of INVSENSOR00039 Healthy Volunteers Needed Advertisement

Confidentiality

Desaturation Validation of INVSENSOR00039 Case Report Form (CRF)

**Post Care Instructions** 

W-9 Request for Taxpayer Identification Number and Certification

Volunteer Payment Form

## 4. LOCATION

Masimo Corporation

Clinical Laboratory

52 Discovery

Irvine, CA 92618



R-TP-20068

## **Desaturation Validation of INVSENSOR00039**



## 5. STUDY POPULATION (\*= PER PHYSICIAN DISCRETION)

#### 5.1. Inclusion Criteria

- Subject is 18-50 years of age.
- Subject weighs a minimum of 110 lbs and no more than 250 lbs unless subject is over 6 feet tall.
- Hemoglobin value is greater than or equal to 11 g/dL.
- Baseline heart rate ≥ 45 bpm and ≤ 85 bpm.
- CO value ≤ 2.0% FCOHb
- Subject has a physical status of ASA I or II (American Society of Anesthesiology Class I; Healthy subjects without any systemic disease at all. American Society of Anesthesiology Class II; subjects with mild systemic disease) as it applies to the systemic disease portion of the classification.
- Blood pressure: Systolic Blood Pressure ≤ 140 mmHg and ≥ 90 mmHg, Diastolic Blood Pressure ≤ 90 mmHg and ≥ 50 mmHg, and if blood pressure is lower than 100/60 subject passes an orthostatic blood pressure test.
- Subject is able to read and communicate in English and understands the study and risks involved.

#### 5.2. Exclusion Criteria

- Subject is pregnant.
- Subject has a BMI > 35 and has been classified as morbidly obese or at an increased risk for participation by a medical professional.
- Subject has a history of fainting (vasovagal), blacking out or losing consciousness during or after blood draw, or has a fear of blood draws.
- Subject smokes one pack of cigarettes or more in one week, and/or the equivalent of e-cigarette liquid, and smokers are not being recruited as indicated in the CSRF.
- Subject has open wounds, inflamed tattoos or piercings, and/oror any visible healing wounds that a medical professional renders them at an increased risk for participation.\*
- Subject has known drug or alcohol abuse and/or use of recreational drugs.
- Subject experiences frequent or severe headaches and/or migraine headaches, migraine auras, altitude sickness, and/or headaches accompanied by visual changes or sensitivity to light or sound.
- Subject has experienced a concussion or head injury with loss of consciousness within the last 12 months.
- Subject has any history of a stroke, myocardial infarction, seizures or heart attack.
- Subject has a chronic bleeding disorder (i.e. hemophilia).
- Subject who has taken anticoagulant medication within the last 30 days (excluding nonsteroidal anti-inflammatory drugs (NSAIDS)).
- Subject has donated blood within the past 4 weeks.
- Subject has Wolff-Parkinson-White Syndrome or Stokes-Adams Syndrome.
- Subject has any symptomatic cardiac dysrhythmia (i.e. atrial fibrillation) and has not received clearance by their physician to participate.
- Subject has a known neurological and/or psychiatric disorder (i.e. schizophrenia, bipolar disorder, Multiple Sclerosis, Huntington's Disease) that interferes with the subject's level of consciousness.
- Subject has taken opioid pain medication 24 hours before the study.
- Subject has any type of infectious disease (i.e. Hepatitis, HIV, Tuberculosis, Flu, Malaria, Measles, etc.).
- Subject is taking medications known to treat any type of infectious disease.\*
- Subject has either signs or history of peripheral ischemia or carpal tunnel syndrome.

# Desaturation Validation of INVSENSOR00039



- Subject has had invasive surgery within the past year- including but not limited to gallbladder, major fracture repairs (involving plates/ screws), jaw surgery, urinary tract surgery, major ENT surgery, joint replacement or gynecological surgeries, heart surgery or thoracic surgery.
- Subject has symptoms of congestion, head cold, flu or other illnesses.
- Subject experiences claustrophobia or has generalized anxiety disorder.
- Subject has been in severe car accident(s) or a similar type of accident(s) requiring hospitalization within the last 12 months.
- Subject has any cancer or history of cancer (not including skin cancer).\*
- Subject has chronic unresolved asthma, lung disease (including COPD) or respiratory disease.
- Subject is allergic to lidocaine, latex, adhesives, or plastic.
- Subject has heart conditions, insulin-dependent Diabetes or uncontrolled hypertension.
- Subject has delivered vaginally, has had a pregnancy terminated, a miscarriage with hospitalization, or had a C-section within the last 6 months.
- Subject intends on participating in any heavy lifting, repetitive movement of their wrist (including
  riding a motorcycle, tennis) or exercise (working out, riding a bike, riding a skate board etc.), or any
  activity that will put additional stress on the wrist within 24 hours following a study that involves an
  arterial line.
- Subject has any medical condition which in the judgment of the investigator and/or medical staff, renders them ineligible for participation in this study or subject is deemed ineligible by the discretion of the investigator/study staff.

## 5.3. Withdrawal of subjects

Subjects must be withdrawn under the following circumstances:

- 5.3.1 The subject withdraws consent.
- 5.3.2 Discretion of investigator, for example:
  - The investigator feels that the subject does not fully comprehend and understand the consent form.



## 5.4. Replacement of subjects

In case a subject is withdrawn from the study, another subject may be recruited.

#### 6. EQUIPMENT AND MATERIALS

Equipment and Materials: All lab analyzers and equipment will be maintained per manufacturer specifications and all study personnel will be trained on the use of relevant equipment. Equivalent equipment and materials to those listed below may be used.

#### Safety Equipment (FDA-Cleared)

Blood pressure monitoring system

R-TP-20068

# **Desaturation Validation of INVSENSOR00039**

- Electrocardiogram (ECG)
- Masimo Pulse Oximeters (Radical-7)
- Masimo Patient Monitoring Platform (Root®)
- Pulse oximeter sensors and cables (Masimo SET, Masimo rainbow, or comparable)
- Medical-grade oxygen tank and mask
- Crash cart

## **Test Devices**

Masimo INVSENSOR00039 sensor – Investigational



#### 7. PROCEDURE

7.1 **SCHEDULE OF ACTIVITIES** 



R-TP-20068

# **Desaturation Validation of INVSENSOR00039**



## 7.2. RECRUITMENT AND PRESCREENING

Subjects will be recruited using IRB-approved advertisements. Subjects may be referred to the study by previous subjects. Subjects are contacted via phone call to conduct a prescreening interview to determine their initial eligibility for the study. Potential eligible subjects are scheduled for a study visit to the clinical laboratory.

#### 7.3 CONSENTING AND SCREENING

Study staff will discuss the informed consent process and the study with the potential subjects. The subjects will be provided with enough time to read and understand the informed consent document and their questions will be answered by study staff prior to the subject signing the informed consent form. No study related activities will be conducted until consent is signed.

Subjects may be asked to provide a copy of their valid government photo ID and/or Social Security Number (SSN) card to verify subject identity. The copies of these forms of identification will be stored along with the subject's consent. The confidentiality and retention of these documents will be protected to the extent provided and required by law.

Subjects will be asked a brief series of health questions to ensure their eligibility for this study. Subjects who do not meet the inclusion and exclusion criteria will not be eligible to participate in the study.

Subject demographic information including age, sex, skin tone, ethnicity, height and weight will be collected. These may be recorded for data analysis and/or subject safety monitoring purposes.

In addition, a medical history will be recorded after the initial screening questionnaire.

Pre-procedure vital signs will be recorded for subject safety monitoring. Spikes in blood pressure and heart rate can be expected during line placement, needle sticks, blood draws etc. and may also be attributed to anxiety/nervousness relating to a new environment. Only the initial recorded blood pressure and/or heart rate determines a subject's qualification for the study.

A physician will perform an orthostatic blood pressure test on subjects whose initial blood pressure is lower than 100/60. The orthostatic blood pressure test will start with the physician taking the subject's blood pressure while they are lying in supine position. The subject will then stand up for 30 seconds and a second blood pressure measurement will be taken. The subject's blood pressure will need to stay above 90/50 to meet inclusion criteria for the study.

Female subjects will be required to take a pregnancy test. Results will be noted in study documentation. If the pregnancy test is positive, the subject will be notified and removed from the study.

A venous sample will be obtained via needle stick or by placement of an IV and analyzed to verify that the subject meets the inclusion criteria for hemoglobin level and HbCO. The subject will be excluded from the study if the values from the blood draw fall outside the ranges stated in the inclusion criteria.

Subjects may have a blanket placed on them for their comfort.

R-TP-20068

## Desaturation Validation of INVSENSOR00039

Subjects may be offered a snack (e.g., granola bar) and/or beverage (e.g., water, juice) due to the amount of time their involvement in this study may take.

#### 7.4. PROCEDURE

The subject will be seated and/or lying in supine position and should refrain from excessive movement during the study.

If accepted into the study, standard noninvasive monitors will be placed on the subject, including ECG, blood pressure, and a reference pulse oximeter (may not be recorded automatically depending on the protocol, this may be recorded manually by medical staff) This is assessed for subject monitoring only.

Proprietary Masimo data collection software will be used to verify all oximeters are reading. If not, proper sensor positioning will be checked and sensors may be repositioned, as needed.



A peripheral venous line will be placed in the subject's hand or arm. This line may be used for the qualifying venous blood draw and for safety or clinical intervention required during the study.

Local anesthetics such as lidocaine, ethyl chloride spray, or Pain Ease skin refrigerant spray may be used in the event that an IV is placed to numb the site. Subjects will be given the option to have lidocaine or numbing spray be used during IV placement for the purpose of making catheter placement more comfortable for the subjects.



Upon successful placement of the sensors and the subject's indication that they are comfortable, a baseline set of blood samples will be obtained.



in a controlled manner to lower the subject's blood oxygen saturation. The lowest targeted value

R-TP-20068

## **Desaturation Validation of INVSENSOR00039**

| | ensure that levels are within the targeted oxygen saturation range and to minimize time that the subject may drop below the targeted range. Note: At any point in the study, if the subject feels uncomfortable, the subject will be given 100% oxygen through either the mouthpiece or a supplemental mask. |
|---|---|
| | The study will end with several minutes at a FiO $_2$ greater than room air (>21%) to help the subject re-saturate after the procedures. |
| | If at any point the subject is uncomfortable with the study, the study will be stopped. |
| 7.5 | END OF STUDY PROCEDURE |
| | At the conclusion of the procedure, the sensors/devices, IV(s), will be removed. A set of post-study vitals will be obtained and recorded on the case report form for safety purposes. The subject will be allowed to leave after medical personnel determine it is safe to do so. |
| | The total procedure time will be approximately |
| | All subjects will be encouraged to remain in the study area until they feel fit to leave; subjects should feel safe and able before returning to work directly after participation in the study. |
| | Study staff may take to verify the subjects blood values are within normal range (eg. pH, Glucose, etc.) |
| | Subjects will be given instructions on wound care. All subjects will be instructed to contact the principal investigator or study staff in the event of any potential complication. |
| | Subjects will be paid for their time. |
| | After the study has ended subjects will be offered a snack (eg. Granola bar) and something to drink (eg. water or juice). Subjects are asked to consume food and/or liquid prior to leaving the clinical lab area for their safety due to study procedures such as blood removal and line placement. Subjects may also be asked to wait in the clinical lab or lobby waiting area leaving to allow for their body to continue adjusting after the study has completed. |

## 7.6 RE-CONTACTING SUBJECTS

If the subject fails to provide proper documentation on their individual consent form for any study, Masimo has the right to re-contact the subject and ask them to return to the clinical lab in order to properly complete the consent form or subject bill of rights. Subject will be compensated for travel.

The subject will also fill out other study documents. These documents aid in the collection of data, tracking subject count, etc. If the subject fails to provide proper documentation on other documents, Masimo has the right to re-contact the subject and ask them to return to the clinical lab in order to properly complete these documents if seen as necessary by study staff.

The subject will be re-contacted via phone or email and be asked to return as soon as possible.

## **Desaturation Validation of INVSENSOR00039**



For validation studies, acceptance criteria is determined by Masimo specifications for each design.

- 9. SAMPLE SIZE JUSTIFICATION AND DATA ANALYSIS PROCEDURE TO BE USED
  - 9.1. Sample size determination



- 9.2. Statistical Analysis
  - a. Exclusion

The following data exclusion criteria will be applied before data analysis:



b. Accuracy calculations

Accuracy will be reported as the A<sub>RMS</sub> using the following equation:

$$Bias = \frac{1}{n} \sum_{i=1}^{n} (Sp02 - Sa02)$$

$$Precision = \sqrt{\frac{\sum_{i=1}^{n} ((Sp02 - Sa02) - Bias)^{2}}{n}}$$

$$A_{RMS} = \sqrt{\frac{\sum_{i=1}^{n} (Sp02 - Sa02)^{2}}{n}}$$

R-TP-20068

## Desaturation Validation of INVSENSOR00039

9.3. The A<sub>RMS</sub> and precision values will be adjusted



9.4. Measures taken to minimize/avoid bias:

9.3.1

9.5. Expected drop out rates

Subjects may not complete the study for various reasons, such as screen failure, unable to complete desaturation criteria, unable to have intravenous or arterial line placed.

#### 10. ADVERSE EVENTS

Definitions:

<u>Adverse event</u>: Any untoward medical occurrence in a subjects, users or other persons, whether or not related to the medical device under study.

<u>Device-related adverse event</u>: Adverse event related to, associated with, or caused by, the use of a medical device under study, including but not limited to events that may have been attributed to the device because of device failure or malfunction, improper or inadequate design, manufacture or user error.

<u>Device deficiency</u>: Inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety or performance. Device deficiencies include malfunctions, use errors and inadequate labeling.

Device deficiencies will be reported according to department procedures.

<u>Serious adverse event</u>: Adverse event that: a) led to death, b) led to serious deterioration in the health of the subject, that resulted in: (i) a life-threatening illness or injury, (ii) a persistent or significant impairment of a body structure or a body function, (iii) in-patient or prolonged hospitalization, or (iv) medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function, or c) led to fetal distress, fetal death or a congenital abnormality or birth defect. NOTE: Planned hospitalization for a pre-existing condition, or a procedure required by the clinical investigational plan, without serious deterioration in health, is not considered a serious adverse event.

All adverse events, including inter-current illnesses will be reported and documented as described below.

#### 10.1. Adverse Events

All adverse events that occur during the study shall be recorded on the Case Report Form even if the investigator/study staff assess the adverse event as unlikely to be causally related to the test device or study procedures.

#### 10.2. Serious Adverse Events

The investigator/study staff shall promptly report both serious adverse events and unanticipated adverse device effects to the sponsor within 48 hours. All serious adverse events will also be reported to the IRB per IRB reporting requirements.

At the time of discharge from the study, any unresolved serious adverse event(s) will be followed up by the investigator/study staff until the event(s) are resolved, stabilized or the patient is lost to

R-TP-20068

## Desaturation Validation of INVSENSOR00039

follow-up or the adverse event is otherwise explained. The investigator and/or study staff will also instruct the subject to report any subsequent events occurring in the next 30 days, which the subject or the subject's physician believes might reasonably be regarded as caused by or have a reasonable possibility of being caused by the test device or procedures involved in the study.

## 10.3. Unanticipated Problems

Any unanticipated problem involving subjects will be reported to the IRB, such as protocol violations or deviations as required by the IRB reporting procedures.

## 11. SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS

- 11.1 Measures Taken to Protect the Rights and Welfare of Subjects
  - 11.1.1 All subjects will be monitored closely throughout the study.
  - 11.1.2 The following measures will be taken to ensure the confidentiality of the subjects:
    - 11.1.2.1 A code (identification) number for each subject will be kept on file.
    - 11.1.2.2 Only their corresponding identification number will identify subjects.
    - 11.1.2.3 Access to identifying documents (IC, SSN, photo ID) and data will only be made to the principal investigators in the study and study staff.
    - 11.1.2.4 The confidentiality and retention of these documents will be protected to the extent provided and required by the law.
- 11.2 Vulnerable Populations



11.2.2 Economically disadvantaged or unemployed and educationally disadvantaged.

Reasonable compensation will be provided for economically disadvantaged subjects to eliminate possibility of undue influence due to financial incentive. Educationally disadvantaged subjects will be provided ample time to ask questions and comprehend information.

- 11.3 Documents and Database
  - 11.3.1 Documents will be kept after the specific product/tested for is no longer being made. If destroyed, these documents will be shredded and done by a certified company used for destroying medical and clinical data.

R-TP-20068

## **Desaturation Validation of INVSENSOR00039**



12.1 Receipt of Study Device

Upon receipt of the study device supplies, an inventory must be performed and the device accountability log filled out and signed by the person accepting the shipment. It is important that the designated study staff counts and verifies that the shipment contains all the items noted in the shipment inventory. Any damaged or unusable study devices in a given shipment will be documented in the study files.

12.2 Use of Study Device

Use of devices and sensors will be documented on Case Report Forms for each subject.

12.3 Return or Destruction of Study Device

At the completion of the study, there will be a final reconciliation of study devices and sensors shipped, devices/sensors used, and devices/sensors remaining. This reconciliation will be logged on the device accountability log. Any discrepancies noted will be investigated, resolved, and documented prior to return or destruction of unused study devices. Devices destroyed on site will only be upon written instruction from the sponsor and will be documented in the study files.

## 13. RISKS AND BENEFITS

- 13.1. Benefits: There will be no benefit to the subject. Other possible benefits would be to society as a whole. Evaluation of the accuracy of this new device could enable healthcare workers to more appropriately treat potentially life threatening conditions.
- 13.2. Device Risks: The noninvasive devices used in this study are similar in technology and design to some commercially available pulse oximeters and other non-invasive devices and hence have the same risks. Pulse oximeters and other non-invasive devices are commonly used and are considered to be minimal risk. There is an extremely small risk of damage to the subject's fingers, or other locations where sensors are placed, from the device including temporary skin irritation or discomfort associated with exposure to the sensor as well as potential temporary mechanical irritation or discomfort. There is a remote, yet possible, risk of a burn from the sensor. In the case of a sensor burn there is the potential for permanent skin damage (scar/discoloration).
- 13.3. Venous Cannulation Risks: swelling, infection, infiltration of fluids/ blood into area surrounding IV, bruising, hematoma, lightheadedness, fainting, feeling flush/warm, feeling nauseated, throwing up, sudden drop in blood pressure/sudden increase in blood pressure, sudden drop in heart rate/sudden increase in heart rate, tingling sensation of face, arms and/or legs, sweating, mouth dryness, damage to the blood vessel and surrounding nerves or tissue.
- 13.4. Arterial Cannulation risks: decreased blood supply, blood clot, embolization, infection, hematoma, damage to the blood vessel and surrounding nerves, tendons or tissue; loss of feeling in hand and/or arm and even the loss of hand due to rare complications of the study.
- 13.5. Blood Draw risks: discomfort is generally associated with needle puncture. The most common complications associated with blood draws and capillary sticks are hematomas or bruising. All blood draws will be performed by qualified personnel. An ACLS certified physician will be in attendance throughout the entire procedure, and the study will be completed under their general supervision.

R-TP-20068

## Desaturation Validation of INVSENSOR00039



- 13.6. Risk From Oxygen Administration: It is expected that some people may experience feelings of claustrophobia or anxiousness from wearing a mouthpiece and/or mask. There are no additional risks associated with high oxygen/oxygen administration for less than 24 hours as long as subjects do not have any cardiac conditions, COPD or any other lung diseases. Subjects' answers on the health questionnaire will help the medical staff decide if they can safely participate in this study; subjects are encouraged to let the study staff know if they have any concerns.
- 13.7. Low Oxygen Concentration Risks: Risks associated with hypoxia include dizziness, shortness of breath, drowsiness, or headache. If or when this occurs, the study can be stopped. There is an extremely small risk of loss of consciousness, damage to vital organs, or death from lack of oxygen. The study shall be stopped by the subject or clinical staff long before this could occur. Other anticipated adverse events that may occur, include but are not limited to: vasovagal (passing out/fainting), lightheadedness, feeling flush/warm, feeling of anxiety, feeling nauseated, throwing up, seizures, sudden drop in blood pressure/sudden increase in blood pressure, sudden drop in heart rate/sudden increase in heart rate, tingling sensation of face, arms and/or legs, sweating, mouth dryness, feeling claustrophobic or anxiousness from wearing a mouthpiece and/or mask. These anticipated adverse events are expected to be temporary.



- 13.10. Risk from Inflicted Knowledge: The risk of inflicted medical knowledge to subjects is negligible since we deidentify all associated sample information including those relevant to our clinical and engineering parameter studies. The monitoring and test results are not examined for diagnostic purposes and do not reflect an attempt to ascertain any subject's medical condition. The attending physician's role during this study is to ensure the safety of the subject during the study. Subjects are informed that these are not diagnostic tools, if observations are made using FDA cleared devices we will refer them to their primary care physician.
- 13.11. Risk From Loss of Confidentiality: Masimo upholds the highest standards to protect hard and electronic data however, a complete promise for confidentiality cannot be guaranteed due to unforeseeable events.
- 13.12. Risk From Additional Testing:

R-TP-20068

## Desaturation Validation of INVSENSOR00039



Within the consent, subjects will agree to permit the company to test the blood sample (or samples) by signing the consent. The test results will be maintained as confidential and will only be used by healthcare professionals for the diagnosis and treatment of the exposed individual as appropriate.

In the case that Masimo needs to contact a subject regarding additional testing they will be contacted by a Masimo employee and medical personnel can be available for further counsel if requested.

The cost for the initial testing and compensation for their time/travel to the testing facility will be the only things paid for by Masimo.

- 13.13. Lidocaine (injection) Risks: Insertion of the Lidocaine may be discomforting and can feel like a slight pinch along with a warm/burning sensation. Other anticipated adverse events that may occur, include but are not limited to: Flushing or redness of the skin, itching skin, small red or purple spots on the skin, unusually warm skin, bruising, bleeding at the application site, swelling, feeling nauseated, dizziness, low blood pressure, and/or tremors. These adverse events are expected to be temporary.
- 13.14. Although not common, it is also possible to have an allergic reaction to injectable lidocaine (e.g., seizures). Subjects should not take part in this study if they are allergic to lidocaine injection or other types of numbing medicine, or if they have a heart rhythm disorder such as Wolff-Parkinson-White Syndrome or Stokes-Adams syndrome. Subjects are instructed to tell the study staff right away if they experience hives; difficulty breathing; swelling of your face, lips, tongue or throat.
- 13.15. Ethyl Chloride (Lidocaine Spray): Ethyl Chloride is a topical anesthetic which is used to prevent pain by cooling the skin. Although unlikely, the anticipated adverse events that may occur, include but are not limited to: changes in skin color (i.e. Flushing or redness of the skin), delayed wound healing, rash, itching and swelling. These adverse events are expected to be temporary.

#### 14. EMERGENCY RESPONSE PLAN FOR MEDICAL EMERGENCIES

The physician and nurse present during the study will be ACLS certified and will respond to any medical emergency involving a subject with the ACLS approved protocol for intervention. A crash cart is on site and full emergency services are within 3 miles.

#### 15. MONITORING PLAN

A separate document for the study monitoring plan will be developed and followed to ensure subject safety and GCP compliance.

#### 16. PROTOCOL DEVIATIONS AND AMENDMENTS

Deviations to the protocol will be documented on the Case Report Form or a separate document. Protocol deviations will be reported to the sponsor and IRB per IRB reporting guidelines.



R-TP-20068

# **Desaturation Validation of INVSENSOR00039**



Modifications to the protocol, informed consent materials, recruitment materials, or any other materials provided to subjects must be reviewed and approved by the IRB.